CLINICAL TRIAL: NCT01330303
Title: Randomized, Two-period, Cross-over, Bioequivalence Study on Tamsulosin Hydrochloride 0,4 mg Prolonged Release Hard Gelatin Capsule Versus SECOTEX® (Tamsulosin Hydrochloride) 0,4 mg Prolonged Release Hard Gelatin Capsule Healthy Male Volunteers Under Fed Conditions
Brief Title: SECOTEX® (Tamsulosin Hydrochloride) Bioequivalence Study Brazil - Fed Admin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 114073
Record Dates: First submitted 2010-08-30; First posted 2011-04-06 (Estimated); Results first posted 2011-04-06 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-06

CONDITIONS: Prostatic Hyperplasia
Keywords: Bioequivalence; Healthy volunteers; tamsulosin hydrochloride; Fed administration
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- tamsulosin - Reference (Active Comparator): Reference drug administration followed by Test drug administration
  Interventions: Drug: Reference formulation; Drug: Test formulation
- tamsulosin - Test (Active Comparator): Test drug administration followed by Reference drug administration
  Interventions: Drug: Reference formulation; Drug: Test formulation

INTERVENTIONS:
Drug: Reference formulation — SECOTEX® (tamsulosin hydrochloride) 0,4 mg (Boehringer Ingelheim)
Drug: Test formulation — tamsulosin hydrochloride 0,4 mg (Synthon BV)

SUMMARY:
It will be an open-label, randomized, laboratory-blind, crossover study with 02 treatments, 02 sequences, and 02 periods, in which the volunteers receive, in each period, the test formulation or the reference formulation, under fed conditions.

DETAILED DESCRIPTION:
It will be an open-label, randomized, laboratory-blind, crossover study with 02 treatments, 02 sequences, and 02 periods, in which the volunteers receive, in each period, the test formulation or the reference formulation, under fed conditions.

The treatment's sequence attributed to each volunteer on the study period is determined by a randomization list, which is generated by PROC PLAN from SAS version 9.1.3 system.

The formulations will be administered as a single oral dose followed by blood collections between, at least, 3 to 5 half-lives. The treatment's periods may obey a minimum interval of 7 half lives between them (period for drug's whole elimination by the organism).

ELIGIBILITY:
EXCLUSION CRITERIA:

* The volunteer has a known hypersensitivity to the study drug (tamsulosin hydrochloride) or to compounds chemically related;
* History or presence of hepatic or gastrointestinal illnesses, or other condition that interferes over the drug's absorption, distribution, excretion or metabolism;
* History of hepatic, renal, pulmonary, gastrointestinal, epileptic, hematologic or psychiatric illness; hypo or hypertension of any etiologic that needs pharmacologic treatment; has history or had myocardial infarction, angina and/or heart insufficiency;
* Non-recommended electrocardiographic findings, according investigator criteria;
* The results of the laboratory exams are out of the values considered as normal according this protocol's rules, unless that they are considered as clinically irrelevant by the investigator;
* Volunteer is a smoker;
* The volunteer ingests more than 5 cups of coffee or tea a day;
* Has history of alcohol or drugs abuse;
* History of serious adverse reactions or hypersensitivity to any drug;
* Use of any regular drug within the 02 weeks that preceded study's initiation or treatment within the 03 previous months, that preceded study's initiation, with any drug that presents toxic, or volunteer consumed inductive drugs and/or enzymatic inhibitor (CYP450 - hepatic), within the 04 weeks that preceded the study's initiation;
* Volunteer was hospitalized for any reason within the 08 weeks of the beginning of the study's first period of treatment and the post study assessment date;
* Participation in any experimental study or ingestion of any experimental drug within the 06 previous months;
* Volunteer consumed alcohol in 48 hours prior to the admission to the study or consumed foods or beverages that contain grapefruit until 07 days previous to each study period.

INCLUSION CRITERIA:

* Male;
* Age between 18 and 50 years;
* Body mass index ≥ 19 and ≤28,5;
* Good health conditions or without significant illness, by judgment of a legally qualified professional, according the rules defined in Protocol, and according the following evaluations: clinical history, pressure and pulse measures, physical and psychological exam, ECG, and additional laboratory exams;
* Capable to understand the study's nature and aim, including the risks and adverse effects and with intention to cooperate with the researcher and to act in compliance with the requirements of the whole assay; this will be confirmed by the Informed Consent's signature.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2009-12-08 (Actual); Primary Completion 2009-12-22 (Actual); Study Completion 2009-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Campinas, São Paulo, Brazil

REFERENCES:
- See also: Results for study 114073 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114073?search=study&search_terms=114073#rs

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Product in Period 1; Reference Product in Period 2: Test product: tamsulosin hydrochloride 0.4 milligrams (mg) prolonged release hard gelatin capsule in Period 1; followed by a 7-day washout period during which no medication was administered; followed by reference product: SECOTEX (tamsulosin hydrochloride) 0.4 mg prolonged release hard gelatin capsule in Period 2
- Reference Product in Period 1; Test Product in Period 2: Reference product: SECOTEX (tamsulosin hydrochloride) 0.4 mg prolonged release hard gelatin capsule in Period 1; followed by a 7-day washout period during which no medication was administered; followed by test product: tamsulosin hydrochloride 0.4 mg prolonged release hard gelatin capsule in Period 2
Period: Period 1
Arm/Group | Test Product in Period 1; Reference Product in Period 2 | Reference Product in Period 1; Test Product in Period 2
Started | 20 | 20
Completed | 19 | 18
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: 7-Day Washout Period
Arm/Group | Test Product in Period 1; Reference Product in Period 2 | Reference Product in Period 1; Test Product in Period 2
Started | 19 | 18
Completed | 19 | 18
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Test Product in Period 1; Reference Product in Period 2 | Reference Product in Period 1; Test Product in Period 2
Started | 19 | 18
Completed | 19 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants Receiving Both Test Product and Reference Product: Participants receiving either test product: tamsulosin hydrochloride 0.4 mg prolonged release hard gelatin capsule in Period 1; followed by reference product: SECOTEX (tamsulosin hydrochloride) 0.4 mg prolonged release hard gelatin capsule in Period 2 or reference product in Period 1 and test product in Period 2
Arm/Group | Participants Receiving Both Test Product and Reference Product
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.20 (7.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 40
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 35
  Mulatto | 3
  Black | 2

OUTCOME MEASURES:

1. Primary Outcome: AUC 0-t
Description: The area under the plot of plasma concentration of drug against time after drug administration is defined as the area under the curve (AUC). The AUC from time 0 (prior to administration of medication) to time t (the time of the last quantifiable concentration) was calculated using the trapezoidal method. This method consists of the sum of the trapezoids' areas, determined by the collection times and their concentrations. The AUC is of particular use in estimating the bioavailability of drugs, by measuring the extent of absorption. ng, nanograms; ml, milliliter.
Time Frame: Day 1 (day that blood collections started) to Day 4 (Period 1) and Days 8 to 11 (Period 2)
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: ng per hour per ml (ng.h/ml)
Groups:
- Test Product: Test product: tamsulosin hydrochloride 0.4 mg prolonged release hard gelatin capsule in both periods
- Reference Product: Reference product: SECOTEX (tamsulosin hydrochloride) 0.4 mg prolonged release hard gelatin capsule in both periods
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 37 | 37
ng per hour per ml (ng.h/ml) | 229.87 (119.88) | 220.85 (98.60)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — This is a bioequivalence study performed to support the register of tamsulosin hydrochloride, produced by Synthon BV, as a branded generic, to be marketed by GlaxoSmithKline Brasil Ltda., according to the requirements of the Brazilian Regulatory Agency - National Agency of Sanitary Surveillance (ANVISA); Ratio T formulation/R formulation = 101.89, 90% CI [94.91 to 109.39] — The ratios between the geometric means of the test (T) and reference (R) formulations were calculated

2. Primary Outcome: AUC0-infinity
Description: The area under the plot of plasma concentration of drug against time after drug administration is defined as the area under the curve (AUC). The AUC from time 0 (prior to administration of medication) to infinity (the time of complete elimination of the drug) was calculated using the trapezoidal method. This method consists of the sum of the trapezoids' areas, determined by the collection times and their concentrations. The AUC is of particular use in estimating the bioavailability of drugs, by measuring the extent of absorption.
Time Frame: Day 1 (day that blood collections started) to Day 4 (Period 1) and Days 8 to 11 (Period 2)
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: ng.h/ml
Groups:
- Reference Product: Reference product: SECOTEX (tamsulosin hydrochloride) 0.4 mg prolonged release hard gelatin capsule in both period
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 37 | 37
ng.h/ml | 237.87 (125.56) | 228.36 (103.28)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio T formulation/R formulation = 101.91, 90% CI [95.00 to 109.33] — The ratios between the geometric means of the test (T) and reference (R) formulations were calculated

3. Primary Outcome: Cmax
Description: Cmax is defined as the maximum or "peak" concentration of a drug observed after its administration. Cmax is one of the parameters of particular use in estimating the bioavailability of drugs, by measuring the total amount of drug absorbed.
Time Frame: Day 1 (day that blood collections started) to Day 4 (Period 1) and Days 8 to 11 (Period 2)
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 37 | 37
ng/ml | 14.06 (6.22) | 14.88 (5.93)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio T formulation/R formulation = 94.04, 90% CI [86.33 to 102.44] — The ratios between the geometric means of the test (T) and reference (R) formulations were calculated

ADVERSE EVENTS:
Arm/Group | Test Product in Period 1; Reference Product in Period 2 | Reference Product in Period 1; Test Product in Period 2
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 6/20 | 8/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product in Period 1; Reference Product in Period 2 (N=20) | Reference Product in Period 1; Test Product in Period 2 (N=20)
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Serum glutamic-pyruvic increased (Investigations) | 0 | 1
Gamma glutamyl transferase increased (Investigations) | 0 | 1
Glucose high (Investigations) | 0 | 1
Serum triglycerides increased (Investigations) | 0 | 2
Serum urea increased (Investigations) | 0 | 3
Serum bilirubin increased (total and indirect) (Investigations) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 0
Postural hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.